CLINICAL TRIAL: NCT07244601
Title: Asessment of Sarcopenia Among Elderly Type 2 Diabetic Patients
Brief Title: Case Control in Sarcopenia Among Elderly Type 2 Diabetic Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Eman Alaa Eldean Mohamed (Other)
Responsible Party: Sponsor-Investigator, Eman Alaa Eldean Mohamed, house office of Internal Medicine, Assiut University, Assiut University
Organization: Assiut University (Other)
Other Study IDs: sarcopenia in elderly diabetic
Record Dates: First submitted 2025-09-23; First posted 2025-11-24 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Diabetic Group: Elderly patients with type 2 diabetes mellitus. Participants will be evaluated for the presence or absence of sarcopenia using muscle ultrasound and clinical criteria.
  Interventions: Diagnostic Test: muscle ultrasound
- Non-Diabetic Group: Elderly patients without diabetes mellitus. Participants will also be assessed for sarcopenia using muscle ultrasound and standard diagnostic criteria.
  Interventions: Diagnostic Test: muscle ultrasound

INTERVENTIONS:
Diagnostic Test: muscle ultrasound — Bedside muscle ultrasound to measure muscle thickness, cross-sectional area and echogenicity

SUMMARY:
1. Assess sarcopenia prevalence in elderly diabetic patients.
2. Evaluate impact of diabetes and its medications on muscle health.
3. detect effect of sacropenia on quality of life on elderly

ELIGIBILITY:
1. Inclusion criteria:

   The study will included all patient ,age ≥ 60 years,diagnosed with type 2 diabetes mellitus at least 5 years duraation according to ADA guideline referance(8) (diabetes can be made if a patient's A1C is 6.5% or higher, their FPG is 126 mg/dL or higher, or their 2-hour plasma glucose during an OGTT is 200 mg/dL or higher. A random plasma glucose of 200 mg/dL or higher, in conjunction with classic symptoms of hyperglycemia, also indicates diabetes)

   ●Able to give informed consent
2. Exclusion criteria:

   * chronic renal disease
   * chronic liver disese
   * Severe cognitive impairment
   * Known neuromuscular diseases affecting mobility
   * malignancy Data of the study will collected over one year duration from 1/2026 _1/2027

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: 1. Inclusion criteria:
     The study will included all patient ,age ≥ 60 years,diagnosed with type 2 diabetes mellitus at least 5 years duraation according to ADA guideline referance(8) (diabetes can be made if a patient's A1C is 6.5% or higher, their FPG is 126 mg/dL or higher, or their 2-hour plasma glucose during an OGTT is 200 mg/dL or higher. A random plasma glucose of 200 mg/dL or higher, in conjunction with classic symptoms of hyperglycemia, also indicates diabetes)
     ●Able to give informed consent
  2. Exclusion criteria:
     * chronic renal disease
     * chronic liver disese
     * Severe cognitive impairment
     * Known neuromuscular diseases affecting mobility
     * malignancy Data of the study will collected over one year duration from 1/2026 _1/2027
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-22 (Estimated); Primary Completion 2027-10-20 (Estimated); Study Completion 2028-10-20 (Estimated)

PRIMARY OUTCOMES:
Prevalence of sarcopenia assessed by muscle ultrasound in elderly diabetic | Within 6 months from the start of recruitment.
  Sarcopenia will be evaluated using muscle ultrasound to measure muscle thickness and echo intensity of the quadriceps muscle. The results will be interpreted according to EWGSOP2 diagnostic criteria, which combine muscle mass and muscle strength parameters
Assessment of muscle strength using handgrip dynamometry | Within 6 months
  Handgrip strength will be measured using a handheld dynamometer, and the average of three attempts for the dominant hand will be recorded.

SECONDARY OUTCOMES:
Quality of life score using the SarQoL questionnaire. | Within 6 months.
  Quality of life related to sarcopenia will be evaluated using the validated SarQoL questionnaire.

REFERENCES:
- [Result] Feng L, Gao Q, Hu K, Wu M, Wang Z, Chen F, Mei F, Zhao L, Ma B. Prevalence and Risk Factors of Sarcopenia in Patients With Diabetes: A Meta-analysis. J Clin Endocrinol Metab. 2022 Apr 19;107(5):1470-1483. doi: 10.1210/clinem/dgab884. PMID 34904651